CLINICAL TRIAL: NCT00076713
Title: Antiphospholipid Syndrome Collaborative Registry (APSCORE)
Acronym: APSCORE
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Robert Roubey, MD, Associate Professor, University of North Carolina, Chapel Hill
Other Study IDs: NIAMS-099; N01AR002248-000 (NIH)
Record Dates: First submitted 2004-02-02; First posted 2004-02-03 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, genomic DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Antiphospholipid Syndrome (APS) is an autoimmune disorder in which the body recognizes certain normal components of blood and/or cell membranes as foreign substances and produces antibodies against them. Patients with these antibodies may experience miscarriages and blood clotting disorders, including heart attacks and strokes. APS may occur in people with systemic lupus erythematosus and other autoimmune diseases, or in otherwise healthy individuals.

The Antiphospholipid Syndrome Collaborative Registry (APSCORE) is a national registry and tissue repository for patients with APS. This registry will collect clinical information and blood samples from people with APS.

DETAILED DESCRIPTION:
Registry participants will have a blood sample drawn and will be interviewed about their medical histories. Participants will be asked to return for a follow-up visit after two years. Clinical, demographic, and laboratory data will be collected. Registry resources will be made available to researchers and medical practitioners to support a broad range of research on the causes, diagnosis, mechanisms, and treatment of APS.

The University of North Carolina at Chapel Hill is the coordinating center and an enrollment site for the registry. There are seven other enrollment sites: Ball Memorial Hospital, Muncie, IN; Duke University, Durham, NC; Hospital for Special Surgery, New York, NY; Johns Hopkins University, Baltimore, MD; Morehouse School of Medicine, Atlanta, GA; University of Texas Health Science Center, San Antonio, TX; and University of Utah Health Science Center, Salt Lake City, UT.

ELIGIBILITY:
Inclusion Criteria:

* Antiphospholipid antibodies with or without associated clinical manifestations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specialty and subspecialty clinics
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2000-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Hospital for Special Surgery, Weill-Cornell University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Health Science Center, Salt Lake City, Utah

REFERENCES:
- [Background] Roubey RA. New approaches to prevention of thrombosis in the antiphospholipid syndrome: hopes, trials, and tribulations. Arthritis Rheum. 2003 Nov;48(11):3004-8. doi: 10.1002/art.11332. No abstract available. PMID 14613259
- See also: Click here for the APSCORE Web site. — http://www.aboutus.org/Apscore.org